CLINICAL TRIAL: NCT06182046
Title: The Effect of BOSU Ball Balance Exercises Added to Complete Decongestive Treatment on Static and Dynamic Balance in Breast Cancer-associated Lymphedema.
Brief Title: Effect of BOSU Exercises Added to Complete Decongestive Treatment on Balance in Breast Cancer-associated Lymphedema.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oya Topuz (Other)
Responsible Party: Sponsor-Investigator, Oya Topuz, Clinical Professor, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PamukkaleU-Karaköseli-001
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: BOSU Ball; Lymphedema; Balance
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Balance exercise with BOSU Ball added to complete decongestive treatment (Experimental): Complete decongestive treatment program consists of manual lymph drainage, multi-layer bandaging, skin/nail care and exercise treatments. The treatment will last 45 minutes/session, 5 sessions/week and 3 weeks. Patients in the intervention group will also receive balance exercises with a BOSU ball. These exercises will be performed in 2 sets, 5 days a week for 3 weeks. Each set will last 15 minutes. It will take 15 sessions in total. These exercises include 10 balance exercise movements performed on a bosu ball.
  Interventions: Procedure: Complete decongestive treatment program; Procedure: Balance exercises
- Active Control group: Complete decongestive treatment (Active Comparator): Patients in this group will receive only a complete decongestive treatment program consisting manual lymph drainage, multilayer bandaging, skin/nail care, and exercise treatments. The treatment will last 45 minutes/session, 5 sessions/week and 3 weeks.
  Interventions: Procedure: Complete decongestive treatment program

INTERVENTIONS:
Procedure: Complete decongestive treatment program — It consists of manual lymph drainage, multi-layer bandaging, skin/nail care and exercise treatments. The treatment will last 45 minutes/session, 5 sessions/week and 3 weeks.
Procedure: Balance exercises — These exercises will be performed in 2 sets, 5 days a week for 3 weeks. Each set will last 15 minutes. It will take 15 sessions in total. These exercises include 10 balance exercise movements performed on a bosu ball.
  Arms: Intervention group: Balance exercise with BOSU Ball added to complete decongestive treatment

SUMMARY:
The aim of the study is to investigate the effect of balance exercises performed with the BOSU ball added to complete decongestive treatment on static and dynamic balance in patients with breast cancer-related lymphedema.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. The patients who had unilateral breast cancer-associated lymphedema according to the 2020 diagnostic criteria of the International Society of Lymphology for at least six months and met the inclusion and exclusion criteria will be randomly divided into 2 groups.

The trial will be carried out at Pamukkale University Department of Physical Medicine and Rehabilitation PAUTERM between December 2023 and June 2025. The local ethics committee approved the study. All women will be informed about the purpose and content of the study and all women will sign written consent to participate in the study.

Group1: Group receiving balance exercise with BOSU Ball added to complete decongestive treatment (Intervention group) Complete decongestive treatment program consists of manual lymph drainage, multi-layer bandaging, skin/nail care and exercise treatments. The treatment will last 45 minutes/session, 5 sessions/week and 3 weeks. Patients in the intervention group will also receive balance exercises with a BOSU ball. These exercises will be performed in 2 sets, 5 days a week for 3 weeks. Each set will last 15 minutes. It will take 15 sessions in total. These exercises include 10 balance exercise movements performed on a bosu ball.

Group 2: Group receiving complete decongestive treatment (Active control group) Patients in this group will receive only a complete decongestive treatment program consisting manual lymph drainage, multilayer bandaging, skin/nail care, and exercise treatments. The treatment will last 45 minutes/session, 5 sessions/week and 3 weeks.

All patients will be evaluated with the following evaluation parameters before the treatment and at the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Patients aged 18-65 years
* Having a history of unilateral mastectomy and lymph node dissection at least one year ago due to breast cancer diagnosis.
* Having unilateral breast cancer-related upper extremity lymphedema (>20% volume difference between the two upper extremities) according to the diagnostic criteria of the - International Society of Lymphology (Committee 2020) for at least six months.
* Not having received lymphedema treatment or exercise therapy for the last six months
* Completing breast cancer primary treatment at least 6 months ago (except hormone therapy/aromatase inhibitors)

Exclusion Criteria:

* Bilateral breast cancer
* Bilateral axillary lymph node dissection
* Metastatic breast cancer
* Receiving ongoing radiotherapy or chemotherapy
* Primary or bilateral lymphedema
* Having active cancer
* Presence of stage 3 lymphedema
* Uncontrolled serious systemic disease (cardiopulmonary diseases, arterial or venous diseases, renal dysfunction, uncontrolled hypertension or hypotension).
* Active or previous infection in the last 3 months (cellulitis, lymphangitis)
* Presence of open wounds
* Having any problems that may affect balance (vestibular, visual, neurological or orthopedic diseases)
* Using medications that may affect body fluid and electrolyte balance (diuretics, etc.).
* Individuals with serious mental and sensory problems
* History of spine surgery in the last 6 months
* Being pregnant
* Body mass index >40 kg/m2

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Static balance measurements | 1 day before rehabilitation
  The TecnoBody Prokin 252 system was used to assess balance in the standing position for all participants. This equipment provides data on the center of pressure path length and the area over which the center of pressure moves. Smaller values indicate greater stability and balance ability in the lower extremities.
Static balance measurements | 3 weeks after the start of rehabilitation
  The TecnoBody Prokin 252 system was used to assess balance in the standing position for all participants. This equipment provides data on the center of pressure path length and the area over which the center of pressure moves. Smaller values indicate greater stability and balance ability in the lower extremities.
Dynamic balance measurements | 1 day before rehabilitation
  The TecnoBody Prokin 252 system was used to assess balance in the standing position for all participants. This equipment provides data on the average track error and stability index.
Dynamic balance measurements | 3 weeks after the start of rehabilitation
  The TecnoBody Prokin 252 system was used to assess balance in the standing position for all participants. This equipment provides data on the average track error and stability index.

SECONDARY OUTCOMES:
Arm circumference measurements | 1 day before rehabilitation
  Arm-hand circumference measurements will be made with a tape measure at four points: metacarpal circumference, wrist, 10 cm below the lateral epicondyle and 15 cm above the lateral epicondyle. The measurement will be made on both upper extremities and the difference between them will be recorded.
Arm circumference measurements | 3 weeks after the start of rehabilitation
  Arm-hand circumference measurements will be made with a tape measure at four points: metacarpal circumference, wrist, 10 cm below the lateral epicondyle and 15 cm above the lateral epicondyle. The measurement will be made on both upper extremities and the difference between them will be recorded.
Arm volumetric measurements | 1 day before rehabilitation
  Arm-hand volume measurements will be made with the help of a water displacement volumeter. After placing a mark 15 cm below the acromioclavicular joint from the anterior on both arms of the patients, they will be dipped into the volumeter one by one up to this level and the overflowing water will be measured.
Arm volumetric measurements | 3 weeks after the start of rehabilitation
  Arm-hand volume measurements will be made with the help of a water displacement volumeter. After placing a mark 15 cm below the acromioclavicular joint from the anterior on both arms of the patients, they will be dipped into the volumeter one by one up to this level and the overflowing water will be measured.
Fall Activity Scale | 1 day before rehabilitation
  It is a 10-item scale. Each question is given a score between 1 (not completely safe) and 10 (very safe), with the total score ranging from 0 to 100. As the score increases, the fear of falling decreases.
Fall Activity Scale | 3 weeks after the start of rehabilitation
  It is a 10-item scale. Each question is given a score between 1 (not completely safe) and 10 (very safe), with the total score ranging from 0 to 100. As the score increases, the fear of falling decreases.
Tampa Kinesiophobia Scale | 1 day before rehabilitation
  It is a checklist of 17 questions. 4-point Likert scoring (1 = Strongly disagree, 4 = Completely agree) is used in the scale. The person receives a total score between 17-68. A high score on the scale indicates that the person has a high level of kinesiophobia.
Tampa Kinesiophobia Scale | 3 weeks after the start of rehabilitation
  It is a checklist of 17 questions. 4-point Likert scoring (1 = Strongly disagree, 4 = Completely agree) is used in the scale. The person receives a total score between 17-68. A high score on the scale indicates that the person has a high level of kinesiophobia.
Fullerton Advanced Balance Scale | 1 day before rehabilitation
  The FAB scale was developed to assess subtle changes in many dimensions of balance. This performance-based scale consists of 10 test items that assess functional balance status in older people. Each test item is scored using a scale of 0-4. The person receives a total score between 0-40. Higher scores indicate better balance ability.
Fullerton Advanced Balance Scale | 3 weeks after the start of rehabilitation
  The FAB scale was developed to assess subtle changes in many dimensions of balance. This performance-based scale consists of 10 test items that assess functional balance status in older people. Each test item is scored using a scale of 0-4. The person receives a total score between 0-40. Higher scores indicate better balance ability.
Timed Up and Go Test | 1 day before rehabilitation
  It is a balance test commonly used to examine functional mobility in community-dwelling, frail older adults. The test requires the subject to stand, walk 3 m, turn and walk backwards, and sit down. Older adults who can complete the task in less than 20 seconds have better balance. In contrast, older adults who require 30 seconds or more to complete the task have worse balance.
Timed Up and Go Test | 3 weeks after the start of rehabilitation
  It is a balance test commonly used to examine functional mobility in community-dwelling, frail older adults. The test requires the subject to stand, walk 3 m, turn and walk backwards, and sit down. Older adults who can complete the task in less than 20 seconds have better balance. In contrast, older adults who require 30 seconds or more to complete the task have worse balance.
Quality of Life Measurement ULL-27 | 1 day before rehabilitation
  ULL-27 quality of life questionnaire, developed specifically for upper extremity lymphedema patients. The scale has physical, psychological and social dimensions. It consists of 27 questions. A high score on the scale indicates that lymphedema negatively affects the quality of life.
Quality of Life Measurement ULL-27 | 3 weeks after the start of rehabilitation
  ULL-27 quality of life questionnaire, developed specifically for upper extremity lymphedema patients. The scale has physical, psychological and social dimensions. It consists of 27 questions. A high score on the scale indicates that lymphedema negatively affects the quality of life.
Hospital Anxiety and Depression Scale | 1 day before rehabilitation
  The scale is used to determine the risk of anxiety and depression in the patient and to measure its level and change in severity. The scale consists of a total of 14 questions. The items in the scale are evaluated on a 4-point Likert scale and are based on a scoring system between 0-3. According to the scoring, 0-1 is considered as not sick, 2 is considered as borderline sick, and 2-3 is considered as seriously ill. The total scores of the subscales are obtained by adding these item scores.
Hospital Anxiety and Depression Scale | 3 weeks after the start of rehabilitation
  The scale is used to determine the risk of anxiety and depression in the patient and to measure its level and change in severity. The scale consists of a total of 14 questions. The items in the scale are evaluated on a 4-point Likert scale and are based on a scoring system between 0-3. According to the scoring, 0-1 is considered as not sick, 2 is considered as borderline sick, and 2-3 is considered as seriously ill. The total scores of the subscales are obtained by adding these item scores.

CONTACTS AND LOCATIONS:
Overall Officials: Oya Topuz, Study Director — Pamukkale University

IPD SHARING:
Plan to Share IPD: No